CLINICAL TRIAL: NCT06705725
Title: Phase I Clinical Study of CBG002 CAR-T Cell in Treatment of Relapsed/refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Carbiogene Therapeutics Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRKBY-102c
Record Dates: First submitted 2024-10-23; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CBG002 CAR-T Cell Suspension (Experimental): Single dose of CAR+ T cells will be infused, and classic "3+3" dose escalation will be applied.
  Interventions: Drug: CBG002 CAR-T Cell Suspension

INTERVENTIONS:
Drug: CBG002 CAR-T Cell Suspension — Single dose of CAR+ T cells will be infused, and classic "3+3" dose escalation will be applied.

SUMMARY:
This is a single arm study to evaluate the efficacy and safety of BCMA-targeted CAR-T cells therapy for patients with relapsed/refractory Multiple Myeloma.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old≤ subjects < 75 years old, all genders;
* Patients volunteered to participate in the study, and they or their legal guardians signed informed consent form (ICF);
* According to the diagnostic criteria of the "The Guidelines for Diagnosis and Treatment of Multiple Myeloma in China (2022)", patients with multiple myeloma are clearly diagnosed;
* Patients without indications for hematopoietic stem cell transplantation；
* Meet the definition criteria of relapsed or refractory multiple myeloma. Patients failed at least 3-line of anti-multiple myeloma therapy have at least 2 complete treatment cycles per line, unless the best response to the therapy was recorded as disease progression; Must have a record of disease progression during or within 12 months after the last treatment;
* Applicable only in the dose expansion phase: the surface BCMA positive percentage of plasma cells of bone marrow samples by flow cytometry is ≥ 50 %;
* Patient has one or more measurable multiple myeloma lesions；
* Patients must have appropriate organ function;
* Patients had no contraindications to peripheral blood mononuclear cell collection;
* ECOG score 0-2;
* Expected survival ≥ 12 weeks;
* Female subjects of childbearing potential must have a negative blood pregnancy test within 7 days prior to cell therapy and not be lactating.

Exclusion Criteria:

* Have a history of allergies to cyclophosphamide, fludarabine, or any component of the cell product;
* Severe cardiovascular and cerebrovascular diseases;
* Severe comorbidities or diseases that the researchers believe will put the patients at inappropriate risk or interfere with the study;
* Have a history of allogeneic hematopoietic stem cell transplantation, or received autologous hematopoietic stem cell transplantation (ASCT) within 12 weeks prior to signing the ICF;
* Central nervous system (CNS) involvement or symptoms of CNS involvement or CNS metastases;
* Stroke or seizure occurred within 6 months prior to signing the ICF;
* Previous plasma cell leukemia;
* Multiple myeloma with extramedullary lesions;
* Previous or screening examination showing amyloidosis;
* Malignant tumor cells with T cell origin revealed by previous pathological examination;
* Having autoimmune disease, immunodeficiency or other disease that requires immunosuppressant therapy;
* Within 5 years prior to signing the ICF, patients with malignancies other than multiple myeloma;
* Uncontrolled active infection;
* Systemic disease judged by the investigator to be unstable;
* More than 5 mg/day of prednisone (or equivalent amounts of other corticosteroids) within 1 week prior to apheresis;
* Have used any CAR-T cell products or other genetically modified T cell therapies;
* Previously received anti-tumor therapy against BCMA targets, including but not limited to antibodies, ADCs or CAR-T;
* History of live vaccination (including live attenuated vaccines) within 4 weeks prior to signing the ICF;
* Any non-hematologic toxicity due to prior therapy that cannot be restored to Grade ≤1 or baseline;
* Patients with grade ≥2 acute graft-versus-host disease (GVHD) (Glucksberg criteria) or extensive chronic GVHD (Seattle criteria) requiring treatment within 4 weeks prior to enrollment, or those who may need to receive anti-GVHD treatment during the trial as judged by the investigator;
* History of alcoholism, drug abuse or mental illness requiring drug intervention within 1 year prior to signing the ICF, which may affect the safety evaluation or compliance as judged by the investigator;
* Other conditions that are considered inappropriate by the investigator to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2024-12-26 (Estimated); Primary Completion 2027-10-25 (Estimated); Study Completion 2028-02-22 (Estimated)

PRIMARY OUTCOMES:
AEs. | 2 years post infusion
  The severity and incidence of treatment-emergent adverse events (TEAEs), treatment-related adverse events (TRAEs), and serious adverse events (SAEs).
DLT | 28 days post infusion
  The Dose Limiting Toxicities (DLTs) are based on drug related adverse events and are specifically defined in study protocol.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 3 months post infusion
  ORR at 3 months post infusion as evaluated by the Investigator
Progression free survival (PFS) | 2 years post infusion
  The time from cell infusion to the first assessment of tumor progression or death from any cause
Overall survival (OS) | 2 years post infusion
  The time from cell infusion to death due to any cause
Duration of remission (DOR) | 2 years post infusion
  The time from the first assessment of the tumor for complete response and above efficacy to the first assessment of disease progression or death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jin, Principal Investigator — Zhejiang University

IPD SHARING:
Plan to Share IPD: No